CLINICAL TRIAL: NCT04874025
Title: Observational Analysis of Treatment With Palbociclib in Patients With Locally Advanced and / or Metastatic RH + / HER 2- Breast Cancer in the First Line of Treatment Within Routine Clinical Practice.
Brief Title: Observational Analysis of Palbociclib Treatment in Patients With First Line Therapy for Locally Advanced and/or Metastatic Breast Cancer
Acronym: PALBOSPAIN
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Fernando Moreno Antón, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: PALBOSPAIN
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer.; Real-world data.; Palbociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ibrance — Observational study of Ibrance 75 mg, 100 mg and 125 mg.

SUMMARY:
Hormone therapy is the primary treatment option for patients with HR+ HER2- breast cancer. Despite its activity, hormone therapy is associated with initial, or more frequently acquired, resistance after exposure to one or more treatment lines.

The combination of palbociclib with hormone therapy significantly increases progression free survival (PFS) compared with hormone therapy in first and second treatment line of HR+ HER2- advanced breast cancer.

These results lead to palbociclib approval by the Food and Drug Administration (FDA) in February 2015, and European Medicines Agency (EMA) approval in November 2016 for first-line treatment of patients with metastatic HR+/HER2-breast cancer in combination with an aromatase inhibitor, and for patients who had previously received hormone therapy in combination with fulvestrant.

In Spain, palbociclib was launched last November 1st, 2017. During this period, approximately 3500 patients have received treatment with Palbociclib, and approximately a half of them in first-line treatment in combination with hormone therapy. The collection of efficacy and toxicity data in the first-line usage in the clinical practice setting is of clinical interest.

ELIGIBILITY:
Inclusion Criteria:

* 1. Documented histologically confirmed breast cancer with ER and/or PgR positive and HER2 negative status.
* 2. Locally advanced or metastatic breast cancer not deemed amenable to curative surgery or curative radiation therapy
* 3. HR+/HER2-

  1. HR+: ER+ or PR+ test before or up to 60 days after MBC diagnosis
  2. HER2-: any HER2 negative test and the absence of a positive test (IHC positive 3+, FISH positive/amplified, Positive NOS) before or up to 60 days after MBC diagnosis
* 4. Female or male patients > 18 years
* 5. Have received at least one dose of palbociclib
* 6. At least 2 document clinical visits
* 7. Treatment with palbociclib should have started from November 2017 to November 2019
* 8. Data from the clinical records should be available.
* 9. Patients must be able to understand and sign informed consent if alive.

Exclusion Criteria:

* 1. Previous treatment with hormonal therapy, targeted therapy or chemotherapy for metastatic disease. Previous anticancer treatment for early breast cancer are allowed.
* 2. Treatment with palbociclib in clinical trial or compassionate use programs
* 3. HER2 + (IHC 3+ or FISH +) tumors in the most recent or previous biopsies
* 4. HR negative tumors in the most recent biopsy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic breast cancer receiving palbociclib in first line in 35 Hospitals from Spain.
Sampling Method: Non-Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Real-world progression free survival (rwPFS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 52 months
  Median time (months) from index date to death, disease progression based on radiology, laboratory evidence, pathology, or clinical assessment until next line therapy, or end of the study, whichever came first, assessed up to 52 months

SECONDARY OUTCOMES:
Overall Survival | Time Frame: From date of index treatment until date of death from any accuse or date of end of study, whichever came first, assessed up to 52 months
  Median time (months) from date of index treatment to date of death. Patients who did not die in the study period are censored at their last date in the study.
Real-world tumor response (rwTR) | From date of index treatment to date of disease progression, date of death, or end of study whichever came first, assessed up to 52 months
  Real-world tumor response is defined as complete response or partial response, based on treating clinician's assessment of radiological evidence for change in burden of disease over the course of treatment
Time to next line of therapy | From date of index treatment to date of next line therapy, date of death, or end of study, whichever came first, assessed up to 52 months
  Median time (months) from date of index treatment to date of next line therapy, date of death, or end of study, whichever came first, assessed up to 52 months
Time to first use of chemotherapy | From date of index treatment to date of first use of chemotherapy, date of death, or end of study, whichever came first, assessed up to 52 months
  Median time (months) from date of index treatment to date of first use of chemotherapy, date of death, or end of study, whichever came first, assessed up to 52 months

CONTACTS AND LOCATIONS:
Locations (36):
- Spain (36):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Univesitario Virgen del Rocío, Seville, Andalusia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Basurto, Bilbao, Basque Country
  - Hospital Universitario Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Guadalajara, Guadalajara, Castilla Y La Mancha
  - Hospital Virgen de la Salud, Toledo, Castilla Y La Mancha
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital Universitario de León, León, Castille and León
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario Vall d´Hebrón, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - ICO Hospitalet, L'Hospitalet de Llobregat, Catalonia
  - Arnau Vilanova Lleida, Lleida, Catalonia
  - Hospital Universitario de Cáceres, Cáceres, Extremadura
  - Hospital Universitario de La Coruña, A Coruña, Galicia
  - Hospital Universitario de Ferrol, Ferrol, Galicia
  - Hospital Cínico Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Elche, Elche, Valencia
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Arnau Vilanova Valencia, Valencia

REFERENCES:
- [Derived] Martinez-Janez N, Ezquerra MB, Manso Sanchez LM, Carrasco FH, Torres AA, Morales S, Ortega PT, Gil VLO, Sampedro T, Conejero RA, Calvo-Martinez L, Galve-Calvo E, Lopez R, de la Pena FA, Lopez-Tarruella S, de Araguiz BAHF, Ruiz LB, Cardenas TM, Chacon JI, Anton FM. First-line therapy with palbociclib in patients with advanced HR+/HER2- breast cancer: The real-life study PALBOSPAIN. Breast Cancer Res Treat. 2024 Jul;206(2):317-328. doi: 10.1007/s10549-024-07287-w. Epub 2024 Apr 1. PMID 38561577